CLINICAL TRIAL: NCT02178826
Title: Nocturnal Enuresis and Rapid Maxillary Expansion - Long Term Effect, Prognostic Factors, Quality of Life and Sleep Quality
Brief Title: Nocturnal Enuresis and Rapid Maxillary Expansion
Acronym: NERME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Collaborators: Örebro County Council (Other Government); Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Ingrid Jönson Ring, Dr, Uppsala University Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LUL-2012/379
Record Dates: First submitted 2014-06-24; First posted 2014-07-01 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Nocturnal Enuresis
Keywords: Nocturnal Enuresis; Rapid Maxillary Expansion; Orthodontics; Polysomnography; Quality of life
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Intervention Model Description: Rapid Maxillary Expansion
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rapid Maxillary Expansion (Experimental): A Rapid Maxillary Expander will be fitted and the palate will be expanded approximately 5mm.
  Interventions: Device: Rapid Maxillary Expansion
- Placebo group (Placebo Comparator): A Sham appliance is fitted and activated for 10-14 days. The patients in this group will after it has been revealed they were randomized into the placebo group have a true Rapid Maxillary Expander fitted and the palate will be expanded approximately 5 mm.
  Interventions: Device: Placebo Appliance

INTERVENTIONS:
Device: Rapid Maxillary Expansion — The Rapid Maxillary Expander will over 10-14 days create a palatal expansion of about 5mm.
  Other Names: Hyrax screw
  Arms: Rapid Maxillary Expansion
Device: Placebo Appliance — The Placebo Appliance looks exactly like the Rapid maxillary Expander but the expansion screw does not work. When the expansion screw is activated it does not create a palatal expansion.
  Other Names: Sham Device
  Arms: Placebo group

SUMMARY:
Nocturnal enuresis (NE) is the involuntary loss of urine that occurs only at night in children aged 5 years or more.

NE is a common problem, affecting about 10% of school children. The prevalence declines with each year of maturity but for some it persists in to adolescents and early adulthood. It can lead to bad self-confidence and low self-esteem, which can have psychosocial consequences.

NE is a multifactorial condition. Three central factors have been identified:

A) Many bedwetting children produce large amounts of urine at night due to a deficiency of the antidiuretic hormone vasopressin.

B) Other children have a lack of inhibition of bladder emptying during sleep. C) Almost all children are deep sleepers with high arousal thresholds. They simply don't wake up when the bladder is full or when it contracts.

There are two well established and evidence based treatments today: the bed-wetting alarm and the pharmacologic treatment desmopressin. The alarm emits a sound when the child wets the bed, which conditions the child to wake up or inhibit bladder emptying. This method is curative for about half of the patients who try this, but relapse occurs. Desmopressin is a synthetic analog of arginine vasopressin and works by decreasing the urine volume at night. About half of the patients become dry with this medication but only as long as they take the medicine. To day, at least 25% of all children with NE do not respond to any of the above treatment.

Rapid maxillary expansion (RME) is a common orthodontic technique to treat patients with a narrow upper jaw. The brace is fitted by an orthodontist, and has a jack-screw, which is activated twice every day for 10-14 days. The procedure is neither painful nor harmful and is not very visible at all.

There are a few reports about children who have become dry after RME treatment. None of them have been randomised or placebo controlled but indicates that quite a few children do become dry after this treatment. A recently carried out study in Sweden show that half of the children became dry after RME treatment. These children were all classed as therapy resistant and had already tried the alarm and medication without success.

The reports are intriguing, but invite the question why a brace would help cure NE? It is likely that sleep and respiration is involved. This study will investigate these children's sleep during the treatment. The trial is a randomised, placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 7-14 years old
* At least 7 wet nights out of 14

Exclusion Criteria:

* Daytime incontinence
* Constipation
* ADHD

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2019-01 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Enuresis frequency | 6 months
  Number of wet night

SECONDARY OUTCOMES:
QoL | Baseline, 6 months
  The validated quality of life questionnaire Paediatric Incontinence Questionnaire
QoL | Baseline, 1 month, 6 months
  The validated quality of life questionnaire OSA 18
Sleep quality | Baseline, 1 month, 6 months
  Polygraphic sleep recordings will be carried out at 3 time points during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid M Jönson Ring, DDS, MSc, Principal Investigator — Uppsala University Hospital; Farhan Bazargani, DDS, PhD, Study Director — Örebro County Council; Tryggve Nevéus, MD, PhD, Study Chair — Uppsala University Hospital
Locations (1):
- Folktandvården Uppsala län, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bower WF, Moore KH, Shepherd RB, Adams RD. The epidemiology of childhood enuresis in Australia. Br J Urol. 1996 Oct;78(4):602-6. doi: 10.1046/j.1464-410x.1996.13618.x. PMID 8944518
- [Background] Neveus T. Nocturnal enuresis-theoretic background and practical guidelines. Pediatr Nephrol. 2011 Aug;26(8):1207-14. doi: 10.1007/s00467-011-1762-8. Epub 2011 Jan 26. PMID 21267599
- [Background] Timms DJ. Rapid maxillary expansion in the treatment of nocturnal enuresis. Angle Orthod. 1990 Fall;60(3):229-33; discussion 234. doi: 10.1043/0003-3219(1990)0602.0.CO;2. PMID 2202238
- [Background] Kurol J, Modin H, Bjerkhoel A. Orthodontic maxillary expansion and its effect on nocturnal enuresis. Angle Orthod. 1998 Jun;68(3):225-32. doi: 10.1043/0003-3219(1998)0682.3.CO;2. PMID 9622759
- [Background] Usumez S, Iseri H, Orhan M, Basciftci FA. Effect of rapid maxillary expansion on nocturnal enuresis. Angle Orthod. 2003 Oct;73(5):532-8. doi: 10.1043/0003-3219(2003)0732.0.CO;2. PMID 14580020
- [Background] Schutz-Fransson U, Kurol J. Rapid maxillary expansion effects on nocturnal enuresis in children: a follow-up study. Angle Orthod. 2008 Mar;78(2):201-8. doi: 10.2319/021407-71.1. PMID 18251602